CLINICAL TRIAL: NCT05227911
Title: The Incidence of Incidental Findings in All Abdominal Surgeries
Brief Title: Incidental Findings in Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Aleppo (Other)
Responsible Party: Principal Investigator, Baraa Shebli, Cardiology Resident, University of Aleppo
Other Study IDs: 14761
Record Dates: First submitted 2022-01-22; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: General Surgery
Keywords: Surgery, General surgery, Incidental findings

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abdominal Surgery Group: Participant undergoing abdominal surgery for any indication
  Interventions: Procedure: Abdominal Surgery

INTERVENTIONS:
Procedure: Abdominal Surgery — Abdominal surgery (laparotomy or laparoscopy) ,which includes proper inspection of the abdominal cavity.

SUMMARY:
Despite the recent advancement in diagnostic modalities, many surgeons experience till this day unexpected findings during the course of surgery. Very few information is available in the medical literature in order to assist the surgeon with the anticipation and preparation to deal with Incidental Findings (IFs). Such valuable information can be of great benefit to the surgeon, as the surgical team can prepare himself better -technically and scientifically- to deal with the common expected IFs. The authors aim to examine the incidence of all IFs in abdominal surgery -laparoscopy or laparotomy- and identify possible associations through a cross-sectional designed study conducted in Aleppo University Hospital - Department of Surgery. The authors collected patients' data who underwent abdominal surgery during the period of the two-consecutive years 2018-2019.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 13 y/o
* patients undergoing laparoscopy or laparotomy that must include a proper inspection of the abdominal cavity

Exclusion Criteria:

* patients aged 13 y/o or less
* patients with incomplete data
* gynecological procedures even if it involves laparotomy or laparoscopy.

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing abdominal surgery whether performed by laparotomy or laparoscopy for any indication, however, the procedure must include proper inspection of the abdominal cavity
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The Incidence of IFs detection | Detection during the time of the procedure itself
  Examine the incidence of the detection of Incidental and unexpected findings in abdominal surgery patients.
IFs identification | Detection during the time of the procedure itself
  The identification of the specific IFs encountered in abdominal surgery patients

SECONDARY OUTCOMES:
The incidence of misdiagnosis events | Detection during the time of the procedure itself
  Examine the incidence of misdiagnosis events in abdominal surgeries
The association between procedure type in IF detection | Detection during the time of the procedure itself
  Examine the association between the type of surgery (laparoscopy or laparotomy) and the detection of IFs.
The association between gender in IF detection | Detection during the time of the procedure itself
  Examine the association between the gender of the patient and the detection of IFs.

CONTACTS AND LOCATIONS:
Locations (1):
- Aleppo University Hospital, Aleppo, Aleppo Provice, Syria

IPD SHARING:
Plan to Share IPD: No
Descriptive information about all sample will be provided with the specific characteristics of patients with encountered IFs